CLINICAL TRIAL: NCT02423044
Title: fMRI Spatial Context and Fear Conditioning
Brief Title: Spatial Context and Fear Learning
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150114; 15-M-0114
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2018-10-30

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; fMRI; Virtual Reality; Shock Threat; Healthy Volunteer
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- Fear is a normal response to a threat. Learning fear can be helpful sometimes. For people with anxiety disorders, fear can be long-lasting and too intense. Researchers want to study how people become fearful of situations. They want to understand how the brain learns when it is helpful to feel fear and when it is not.

Objective:

- To better understand brain processes related to fear and anxiety.

Eligibility:

* Right-handed adults ages 18 50 with generalized anxiety disorder, panic disorder, social anxiety disorder, or post-traumatic stress disorder.
* Right handed volunteers ages 18-50 without psychiatric disorders.
* And free of psychiatric medication for 2 weeks

Design:

* Participants will first be screened under another protocol.
* Participants will play a video game inside a magnetic resonance imaging (MRI) scanner. The scanner is a metal cylinder It is surrounded by a strong magnetic field. Participants will lie on a table that can slide in and out of the scanner. A device called a coil will be placed over the head.
* During the scan, participants may play a virtual reality video game. Game instructions will be explained before they enter the scanner.
* While playing the game, participants will wear 2 electrodes on their fingers. These measure sweat on the skin. They will also have 2 small electrodes attached to the left hand. These can give brief mild electrical shocks.
* Participants will be asked questions when playing the game during the scan.
* Before and after the scan, participants will fill out questionnaires about their emotions. They may complete questionnaires online while at the clinic.

DETAILED DESCRIPTION:
Objective:

To examine the processes involved in distinguishing between threatening and safe conditions, we aim to investigate the neural bases of contextual fear learning using functional magnetic resonance imaging (fMRI). To do this, we will study behavioral, physiological, and brain responses as aversive stimuli are encountered in a virtual environment, and will explore how fear-related responses depend on the surrounding environment. In addition, we will examine how these responses differ in clinical anxiety.

We are interested in studying Pavlovian aversive context conditioning in healthy controls and patients with anxiety disorders. We will examine the extent to which participants learn to discriminate between dangerous and safe virtual contexts, and how this learning maps to the neural networks underlying anxiety and context coding. We expect successful learning of the contextual fear response in healthy controls, as evidenced by differential skin conductance response and neural activation to safe vs. threat context. Accordingly, we anticipate higher neuronal activity in the hippocampus, prefrontal cortex, and amygdala. These findings will be accompanied with increased hippocampus-prefrontal cortex connectivity during approach and exploration of the dangerous context, and increased amygdala activation during anticipation of shock in the dangerous context. Physiologically, SCR will increase in threat context compared to safe context. However, anxious patients are expected to fail to learn to differentiate safe from threat context, exhibiting increased SCR and neural activation in both safe and threat contexts, an index of contextual generalization of fear. Particularly, the lack of contextual fear discrimination in anxious patients will be associated with weaker hippocampal activation to contextual learning. To examine differential context fear conditioning, we will use a virtual reality (VR) paradigm. VR provides an optimal way to probe spatial navigation and simulates context. The VR task presents an outdoor space, which comprises a dangerous (probabilistic electrical shocks) and a safe (no shocks) location. Healthy controls and patients with anxiety disorders will be compared on their physiological and neural reactivity during task performance. Preliminary psychophysiological data suggest that the proposed procedure is an effective way to promote different responses to a safe and dangerous spatial location. Hence, we anticipate that this procedure will allow us to examine brain correlates of differential contextual fear responses in humans and compare them between healthy participants and patients diagnosed with an anxiety disorder.

Study population:

Two study populations, healthy volunteers and patients diagnosed with an anxiety disorder (generalized anxiety disorder (GAD), social anxiety disorder (SAD), panic disorder, and post-traumatic stress disorder) will complete the protocol. Participants will be adult males and females, aged 18 to 50 years.

Design:

This fMRI study will compare performance, physiological and neural measures between healthy adults and patients with anxiety disorders, who perform a threat VR task in the scanner.

The VR task entails navigating in a virtual outdoor environment, which, unbeknownst to the participants is divided into a safe and a dangerous context, which are recognizable by environmental characteristics (e.g., mountain, clouds). The dangerous context is associated with probabilistic shocks, which are never encountered in the safe context. Participants learn about these two contexts as they collect flowers (cues), one at a time, in either context. In the dangerous context, the flowers are associated with 50% chance of a shock

Outcome measures:

The primary outcome measures will be the cerebral fMRI blood-oxygen-level dependent (BOLD) responses to three events: (1) shock anticipation: after collecting the cues (flowers) during anticipation of a potential shock, (2) context exploration: as participants navigate in the threat context or safe context in between trials (which start when a flower appears in the environment), and (3) cue approach: during approach towards the flower, in the threat or safe context. The secondary outcome measures will consist of the changes in psychophysiological responses, such as SCR, heart rate, pupil dilatation, and respiratory rate, which will validate fear responses.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages 18-50
* Subjects able to give their consent
* Right handed
* Patients only: a primary diagnosis of GAD, panic disorder, SAD, or PTSD according to the Structured Clinical Interview for DSM-IV-TR

EXCLUSION CRITERIA:

* Non-English speaking individual
* Any significant medical or neurological problems (e.g. cardiovascular illness, respiratory illness, neurological illness, seizure, etc.)
* High or low blood pressure (SBP>140 or SBP<90; SDP<50 or SDP>90)
* Alcohol/drug abuse in the past year or lifetime alcohol or drug dependence according to the Structured Clinical Interview for DSM-IV-TR
* Medications that act on the central nervous system (e.g., Lorazepam, Codeine) and thus may interfere with the interpretation of study results. Specific exclusionary drug classes include but are not limited to: (opioid analgesics, DA receptor agonists, anticholinergics, MAO inhibitors, COMT inhibitors, as well as any illicit substances)
* Pregnancy or positive pregnancy test
* Neurological syndrome of the wrist (e.g., carpal tunnel syndrome, cubital tunnel syndrome, etc.)
* Positive urine toxicology screen
* IQ <80
* Participants who report getting severe motion sickness, especially by playing video games
* Any medical condition that increases risk for fMRI:

  * Any metal implants (clips, screws, plates, pins, etc) or metal fragments cause by injuries or metal working
  * Any sort of medical implants (aneurysm clips, pacemaker, insulin pump, Hickman line, etc.)
  * Permanent eye liner and tattoos above the neck
  * Patients who have difficulty lying flat on their back for up to 60 min in the scanner
  * Participants who are uncomfortable in small closed spaces (have claustrophobia) and would feel uncomfortable in the MRI machine

Additional Exclusion Criteria for Healthy Volunteers:

* Current or past Axis I psychiatric disorders as identified with the Structured Clinical Interview for DSM-IV-TR, non-patient edition (SCID-np)
* Current use of psychotropic medications (i.e. fluoxetine (Prozac), fluvoxamine (Luvox), sertraline (Zoloft), paroxetine (Paxil), citalopram (Celexa) or escitalopram (Lexapro), etc.).

<TAB>

Additional Exclusion Criteria for Patients:

* Patients who are currently on psychotropic medications. (Patients are required to be free of all psychotropics medication (i.e. fluvoxamine (Luvox), sertraline (Zoloft), paroxetine (Paxil), citalopram (Celexa) or escitalopram (Lexapro), etc.) for 2 weeks, 5 weeks for fluoxetine prior to testing. Patients will not be taken off medications for the purpose of the study)
* Patients will be excluded if they have a current or past history of any psychotic disorder, delirium, dementia, amnestic disorder, cognitive disorder not otherwise specified, any of the pervasive developmental disorders, or mental retardation
* Patients who have a primary diagnosis of major depressive disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2015-04-18; Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
The primary objective is to investigate the neural bases of contextual fear learning measures by the event-related hemodynamic response (fMRI). | 12/29/16

SECONDARY OUTCOMES:
The secondary objective is to see learning of the contextual fear response that will be measured by psychophysiological responses such as SCR, heart rate, pupil dilatation, and breathing. | 12/29/16

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ernst, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Britton JC, Lissek S, Grillon C, Norcross MA, Pine DS. Development of anxiety: the role of threat appraisal and fear learning. Depress Anxiety. 2011 Jan;28(1):5-17. doi: 10.1002/da.20733. Epub 2010 Aug 23. PMID 20734364
- [Background] Huff NC, Zeilinski DJ, Fecteau ME, Brady R, LaBar KS. Human fear conditioning conducted in full immersion 3-dimensional virtual reality. J Vis Exp. 2010 Aug 9;(42):1993. doi: 10.3791/1993. PMID 20736913